CLINICAL TRIAL: NCT00907309
Title: Dental and Medical Office Internet/Intranet Motivational Enhancement Therapy to Reduce Teen Tobacco, Alcohol, and Drug Use
Brief Title: Dental and Medical Office iMET to Reduce Teen Tobacco, Alcohol, and Drug Use
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Collaborators: Cambridge Health Alliance (Other); Tufts Medical Center (Other); Harvard School of Dental Medicine (Other); Fallon Clinic (Industry)
Responsible Party: Principal Investigator, John R Knight, MD, Associate Professor of Pediatrics, Harvard Medical School; Senior Associate in Medicine; Associate in Psychiatry, Director, Center for Adolescent Substance Abuse Research, Boston Children's Hospital, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: iMET RFA-OD-09-003
Record Dates: First submitted 2009-05-20; First posted 2009-05-22 (Estimated); Last update posted 2016-10-07 (Estimated); Status verified 2016-10

CONDITIONS: Use; Tobacco, Harmful; Alcohol Abuse; Drug Abuse
Keywords: alcohol abuse; marijuana abuse; drug abuse; tobacco use; tobacco dependence
MeSH Terms: conditions — Alcoholism; Substance-Related Disorders; Marijuana Abuse; Tobacco Use; Tobacco Use Disorder | interventions — histaminol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Treatment as usual (No Intervention): Participants will receive treatment as usual from their provider.
- iMET (Experimental): Participants will receive the iMET intervention.
  Interventions: Behavioral: iMET
- iMET/TE (Experimental): Participants will receive the iMET intervention and Technological Extenders (TEs).
  Interventions: Behavioral: iMET/TE

INTERVENTIONS:
Behavioral: iMET — Participants will receive the iMET intervention
  Arms: iMET
Behavioral: iMET/TE — Participants will receive the iMET intervention and also receive TEs (Technological Extenders)
  Arms: iMET/TE

SUMMARY:
The purpose of the project is to improve adolescent behavioral counseling services in healthcare settings with a new Internet/Intranet-based Motivational Enhancement Therapy (iMET) intervention that targets the use of tobacco, alcohol, and other drugs.

DETAILED DESCRIPTION:
We have previously developed and tested in a treatment population a promising MET program for alcohol and drug use. We will broaden the MET intervention to also target tobacco use and convert the new materials into a self-administered format.

ELIGIBILITY:
Inclusion Criteria:

* 12-21 years old
* Coming for routine care

Exclusion Criteria:

* Medically or emotionally unstable day of visit
* Already receiving behavioral health services
* Cannot read/understand English
* Will not be available for post-tests

Ages: 12 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 121 (Actual)
Dates: Start 2010-09; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Frequency of tobacco, alcohol, marijuana, and other drug use | 3 months, 6 months

SECONDARY OUTCOMES:
Rates of initiation and cessation of tobacco, alcohol, marijuana and other drug use | 3 months, 6 months

CONTACTS AND LOCATIONS:
Overall Officials: John R. Knight, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Children's Hospital Boston, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Holliday R, Hong B, McColl E, Livingstone-Banks J, Preshaw PM. Interventions for tobacco cessation delivered by dental professionals. Cochrane Database Syst Rev. 2021 Feb 19;2(2):CD005084. doi: 10.1002/14651858.CD005084.pub4. PMID 33605440
- See also: web site of Center for Adolescent Substance Abuse Research at Children's Hospital Boston — http://www.ceasar.org